CLINICAL TRIAL: NCT02663583
Title: Observational Parallel Cohort Study of Intensity-Modulated Proton Therapy (IMPT) or TransOral Robotic Surgery (TORS) for the Treatment of Low-Risk Oropharynx Squamous Cell Carcinoma
Brief Title: Intensity-Modulated Proton Therapy (IMPT) or TransOral Robotic Surgery (TORS) for the Treatment of Low-Risk Oropharynx Squamous Cell
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA15-0744
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cancer of the Mouth; Oropharynx Squamous Cell Carcinoma
Keywords: Oropharynx squamous cell carcinoma; OPSCC; Actigraph accelerometer; MD Anderson Symptom Inventory - Head and Neck module; MDASI-HN; Intensity-Modulated Proton Therapy; IMPT; TransOral Robotic Surgery; TORS; Surveys; Questionnaires
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensity-Modulated Proton Therapy or( IMPT) Group: Symptom questionnaires about symptoms of cancer and how they affect life at work and at home, diet, and speech completed at baseline, every week during IMPT, at 3 months, and at 6 months.
  Dysphagia Inventory questionnaire about how difficult it is to swallow completed at baseline, every week during IMPT, at 3 months, and at 6 months.
  Activity bands given to participant at baseline. Participant wears the band 24 hours a day for 1 week leading up to all study visits.
  Interventions: Behavioral: Symptom Questionnaires; Behavioral: Dysphagia Inventory Questionnaire; Behavioral: Activity Bands
- TransOral Robotic Surgery (TORS) Group: Symptom questionnaires about symptoms of cancer and how they affect life at work and at home, diet, and speech completed at baseline, after TORS, at 3 months, and at 6 months.
  Dysphagia Inventory questionnaire about how difficult it is to swallow completed at baseline, after TORS, at 3 months, and at 6 months.
  Activity bands given to participant at baseline. Participant wears the band 24 hours a day for 1 week leading up to all study visits.
  Interventions: Behavioral: Symptom Questionnaires; Behavioral: Dysphagia Inventory Questionnaire; Behavioral: Activity Bands

INTERVENTIONS:
Behavioral: Symptom Questionnaires — Intensity-Modulated Proton Therapy or( IMPT) Group: Symptom questionnaires about symptoms of cancer and how they affect life at work and at home, diet, and speech completed at baseline, every week during IMPT, at 3 months, and at 6 months.
  TransOral Robotic Surgery (TORS) Group: Symptom questionnaires about symptoms of cancer and how they affect life at work and at home, diet, and speech completed at baseline, after TORS, at 3 months, and at 6 months.
  Other Names: Surveys
Behavioral: Dysphagia Inventory Questionnaire — Intensity-Modulated Proton Therapy or( IMPT) Group: Dysphagia Inventory questionnaire about how difficult it is to swallow completed at baseline, every week during IMPT, at 3 months, and at 6 months.
  TransOral Robotic Surgery (TORS) Group: Dysphagia Inventory questionnaire about how difficult it is to swallow completed at baseline, after TORS, at 3 months, and at 6 months.
  Other Names: Survey
Behavioral: Activity Bands — Activity bands given to participant at baseline. Participant wears the band 24 hours a day for 1 week leading up to all study visits.

SUMMARY:
The goal of this laboratory research study is to learn about symptoms and activity levels of patients with OPSCC that receive IMPT or TORS.

DETAILED DESCRIPTION:
Baseline Visit:

If participant agrees to take part in this study, they will complete the following tests and procedures at their baseline visit. This baseline visit will take place before participant's treatment with IMPT or TORS:

* Participant will complete questionnaires about any symptoms of cancer they may be having and how they affect their daily life at work and at home, their diet, and their speech.
* Participant will complete the Dysphagia Inventory. This is a questionnaire about how difficult it is to swallow.
* The study staff will measure how wide participant can open their jaw to see if their treatment may cause any jaw opening limitations.

It should take about 30 minutes to complete all of the questionnaires.

As part of participant's baseline visit, information below will be collected from their medical record:

* Participant's medical history
* The results of participant's physical exam including their weight and any recent weight loss.
* Any other diseases participant may have and any drugs they are currently taking.
* Participant's current smoking status and smoking history.

Activity Bands:

The study staff will either give participant an activity band at their baseline visit or they will be mailed an activity wristband. Participant will be asked to wear the band 24 hours a day for 1 week leading up to all study visits. The wristband will record how active participant is and how much they sleep. The study staff will show participant how to wear and use the wristband.

Study Visits:

Participant will complete the following study procedures after they complete treatment with either IMPT or TORS, and at 3 and 6 months after that.

* The data from participant's wristband will be collected.
* Participant will complete the same questionnaires they did at baseline.
* At participant's 3 month visit only, the study staff will measure how wide they can open their jaw to see if their treatment may cause any jaw opening limitations.

IMPT patients only:

If participant is receiving IMPT, they will complete the questionnaires they completed at the baseline visit once a week while they are receiving treatment.

Length of Study:

Participant's active participation in this study will be over after the 6 month study visit.

Participant will return the wristband to the study staff after their participation is over. If participant loses or damages the wristband while they are on study, another one will be provided to them at no cost.

This is an investigational study.

Up to 44 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically documented or suspected, previously untreated OPSCC (Clinical Stage I-Va; Tx,0-2, N0-2b) eligible for standard of care single-modality treatment with either IMPT or TORS. Patients with suspected OPSCC must have a diagnosis confirmed prior to treatment per the current clinical standard of care
3. Eastern Cooperative Oncology Group (ECOG) = 0, 1, or 2

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants having treatment with either proton therapy (called Intensity-Modulated Proton Therapy or IMPT) or robotic surgery (called TransOral Robotic Surgery or TORS) at MD Anderson Cancer Center in Houston, Texas.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective Functional Outcome After Treatment with Either Intensity-Modulated Proton Therapy (IMPT) or TransOral Robotic Surgery (TORS) in Participants with Low-Risk Oropharynx Squamous Cell Carcinoma (OPSCC) | 6 months
  Functional outcome measured by using longitudinal digital wristband activity monitoring of study participants.
Objective Functional Outcome After Treatment with Either Intensity-Modulated Proton Therapy (IMPT) or TransOral Robotic Surgery (TORS) in Participants with Low-Risk Oropharynx Squamous Cell Carcinoma (OPSCC) | 6 Months
  Functional outcome measured by using patient-reported outcome (PRO) measures from the M.D. Anderson Symptom Inventory for Head and Neck Cancer (MDADI-HN).

CONTACTS AND LOCATIONS:
Overall Officials: Neil Gross, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org